CLINICAL TRIAL: NCT04033978
Title: Cerebral Impact of Cognitive Remediation for People Suffering From Schizophrenia
Acronym: IMPACTRCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminée
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-A00813-54
Record Dates: First submitted 2019-07-05; First posted 2019-07-26 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive remediation; Jumping to Conclusion
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation; Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: The participants don't know the select group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive remediation arm (Experimental): Participants will be enrolled in a cognitive remediation group. The program will last 10 weeks and be composed of 10 participants. This program is based on strategy learning and its aim is to reduce the jumping to conclusion phenomenon.
  Interventions: Behavioral: Cognitive remediation
- Control group (Active Comparator): Participants will be enrolled in an information control group. They will receive information about psychosocial rehabilitation and recovery process. The program lasts 10 weeks.
  Interventions: Behavioral: psychosocial rehabilitation

INTERVENTIONS:
Behavioral: Cognitive remediation — 10 sessions dealing with emotion recognition, jumping to conclusion, attributional style.program lasts 10 weeks
  Arms: Cognitive remediation arm
Behavioral: psychosocial rehabilitation — 10 sessions dealing psychosocial rehabilitation, neuropsychological evaluation, stigmatization, recovery process and severe mental disorders in general.
  Arms: Control group

SUMMARY:
Neurocognitive deficits are frequent with people suffering from schizophrenia. Unlike positive symptoms, cognitive deficits are not reduced with antipsychotic medication. They can be very disabling, especially for social and professional rehabilitation. Cognitive deficits can concern primary processes such as attention or more integrative processes. Social cognition is also massively altered. As a consequence, decision making is often altered with the presence of the 'jumping to conclusion' (JTC) phenomenon. People that jump to conclusion are making decisions without having the necessary information to be sure of their judgment. In addition, people suffering from schizophrenia also present differences in cerebral activity. For instance, the P300 involved in executive processes appears later and with a smaller amplitude. Many cognitive remediation programs have been created to overcome these deficits. Their efficiency has been proved. However, their effects on cerebral activity have not been studied extensively in literature, especially concerning decision making changes. The present project will use a cognitive remediation program centered on social decision making to test its efficiency on JTC and the potential changes in cerebral activity it can induce. This program, inspired by the SCIT (Social Cognition and Interaction Technique) will be based on 10 sessions (1 each week). Participants will be tested before and after remediation/control group with 3 experimental tasks. Cerebral activity will be measured with an EEG cap. They will also undergo a neuropsychological evaluation and a symptomatology evaluation.

DETAILED DESCRIPTION:
Among cognitive deficits associated to schizophrenia, the jumping to conclusion bias is a frequent consequence of the decision making process alteration. This bias is characterized by a fast decision making when probabilistic judgments would be necessar.

Cognitive remediation aims at reducing the impact of cognitive deficits. The program that will be used in the present study focuses on the jump to conclusion bias. In schizophrenia, the positive impact of programs targeting such a bias, and more generally social cognition, has already been shown in numerous studies. However, despite the fact that jumping to conclusion is one of the main goals of these programs, their effects on decision making are poorly investigated in literature.

The program should impact decision making and reduce the jumping to conclusion bias. The benefits will probably be linked with a change in the P300 signal. They will probably appear earlier and with bigger amplitudes.

ELIGIBILITY:
Inclusion Criteria:

* People suffering from schizophrenia given the DSM-5
* People aged from 18 to 45 years old
* French mother tongue
* Medicated with Aripiprazole
* Medication unchanged in the last month
* Stable symptomatology
* People consenting to the research.

Exclusion Criteria:

* Recent addiction (tabacco excluded)
* Neurologic disorders (vascular disorders, neurodegenerative disorders, infections…)
* Somatic medication having cerebral impact (such as corticoids)
* Pregnant women, guardianship people.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Jumping to the conclusion | 12 weeks
  The primary outcome will be modification before and after intervention of the correct response percentage. It is obtained by measuring the amplitude of the waves P300 and N200 of the electroencephalogram.

SECONDARY OUTCOMES:
Warwick-Edinburg mental well-being (WEMWBS) | 12 weeks
  The outcome measure of mental well-being will be the score of scale modification before and after intervention. It is a questionnaire that includes 14 items.
The positive and the negative symptoms (PANNS) | 12 weeks
  The measure of the cognitive fonctioning will be the modification before and after intervention of the score obtained at the proposed neuropsychological evaluation ( excecutive, attentional and social)

CONTACTS AND LOCATIONS:
Overall Officials: FRANCK Nicolas, Professor, Principal Investigator — CH Le Vinatier
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France